CLINICAL TRIAL: NCT06093815
Title: Prospective, Single Site, Controlled Comparative Study to Identify and Assess Tissue Responses After Injection With Various Biostimulatory Products
Brief Title: Prospective Study to Assess Tissue Responses After Injection With Biostimulatory Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Merz North America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: M900311010
Record Dates: First submitted 2023-10-05; First posted 2023-10-23 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Injection Site Reaction
MeSH Terms: conditions — Injection Site Reaction | interventions — Injections

STUDY DESIGN:
Intervention Model Description: Injections will be in redundant abdominal tissue scheduled to be removed at end of study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Arm 1 (Experimental): Subjects in Arm 1 will receive injections of biostimulatory products (Radiesse, Sculptra, Ellanse, HArmonyCa) at 3 timepoints (six months, three months and two weeks) prior to removal of redundant abdominal tissue.
  Interventions: Device: Injection
- Arm 2 (Experimental): Subjects in Arm 2 will receive injections of 1 of 2 selected biostimulatory products (Radiesse or Sculptra) at 1 timepoint (6 months) prior to removal of redundant abdominal tissue.
  Interventions: Device: Injection

INTERVENTIONS:
Device: Injection — A pre specified amount will be injected in tissue at selected timepoints

SUMMARY:
The objective of this study is to identify and assess in vivo tissue responses after injection with various biostimulatory products at various timepoints. The study will also provide tissue specimens which will be used in a subsequent study.

Safety endpoint: incidence of adverse events.

DETAILED DESCRIPTION:
The objective of this study is to identify and assess tissue responses after injection with various biostimulatory products that are already used in the market and have CE approval. The study will assess in vivo tissue responses and provide tissue specimens which will be used in a subsequent study, under a separate protocol.

Assessments under this protocol will include ultrasound of in vivo tissue.

Safety endpoint: incidence of adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male & females; 22 to 65 years of age.
2. Voluntary participation
3. Ability to comprehend and provide informed consent.
4. Participants agree NOT to use any topical agents or products that will induce skin peeling or change the appearance of the skin in the treatment area, during the study period.
5. Participants agree NOT to undergo any aesthetic treatments that influence the appearance of the skin in the treatment area during the study period.
6. Participants agree NOT to undergo any surgical treatments in the treatment area during the study period.
7. Participants agree NOT to take part in another clinical study or undergo other treatments during the study period.

Exclusion Criteria:

1. Any previous surgery in the abdominal area.
2. Any previous treatment in the abdominal area.
3. Planning to receive treatment of any kind in the abdominal area.
4. Acute inflammatory process and/or infection at the injection site.
5. Treatment of skin area with dermatosis.
6. Eczema, exanthema or open wounds.
7. Previous application of over the counter or prescription, oral or topical, anti-wrinkle or skin enhancer products on the abdominal skin within the past 3 months unless allowed by the study and is continued throughout the study.
8. Any contraindication to treatment with biostimulatory products based on the product's IFU.
9. Previous pregnancy or intending to become pregnant during study participation.
10. Known hypersensitivity to biostimulatory products or any of their formulation ingredients.
11. Allergic reaction to topical and local anesthetics.
12. Currently using anticoagulant therapy.
13. Haemophilia / bleeding disorder.
14. Chemotherapy, radiotherapy or high doses of corticosteroids.
15. Systemic infection (e.g., hepatitis).
16. Uncontrolled diabetes mellitus.
17. Any medical condition that may put the participant at increased risk with exposure to biostimulatory products.
18. Any medication that might modulate the immune response.
19. Any other illness or condition that, in the opinion of the investigator, would mean that study participation was not in the best interest of the prospective participant.
20. Is a female of childbearing potential and not using medically effective birth control or is pregnant or lactating.
21. Any serious disease or disorder (medical or psychiatric) that could, in the opinion of the investigator, interfere with the safe completion of treatment according to this protocol or with study.
22. Injection of local anesthesia into the flap during abdominoplasty surgery.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-09-08 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Ultrasound Analyses | 6 months, 3 months and 2 weeks prior to surgery timepoint(s)
  Ultrasound of injection site tissue analyses (dermal thickness (mm), elastosis (mm) and microvascular formation) by PI at various timepoints

OTHER OUTCOMES:
Safety Assessment | through study completion, an average of 6 months
  Adverse event reporting

CONTACTS AND LOCATIONS:
Overall Officials: Ann P Marx, MD, Study Director — Merz North America, Inc.
Locations (1):
- Ocean Clinic - Av. Ramon y Cajal 7, 29601, Marbella, Spain

IPD SHARING:
Plan to Share IPD: No
individual data will be summarized for analyses